CLINICAL TRIAL: NCT04498975
Title: Exploring Potential Associations Between Rurality and Hopelessness in IHD Patients
Status: Completed | Type: Observational
Sponsor: Dordt University (Other)
Collaborators: Sanford Health (Other); Avera McKennan Hospital & University Health Center (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: Hopelessness-Rurality
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Disease; Mental Health Issue
Keywords: Rurality
MeSH Terms: conditions — Heart Diseases | interventions — Ethnicity; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with IHD: No intervention
  Interventions: Other: Rurality; Ethnicity; Exercise; Hopelessness

INTERVENTIONS:
Other: Rurality; Ethnicity; Exercise; Hopelessness — Observational study exploring rurality, ethnicity, exercise and hopelessness patterns cross-sectionally and longitudinally

SUMMARY:
Hopelessness is associated with 3.4 times increased risk of mortality or nonfatal myocardial infarction in patients with ischemic heart disease (IHD), independent of depression. Hopelessness has been identified in 27-52% of patients with IHD and can persist for up to 12 months after hospital discharge. Hopelessness, a negative outlook and sense of helplessness toward the future, can be a temporary response to an event (state) or a habitual outlook (trait). Hopelessness is associated with decreased physical functioning and lower physical activity (PA) levels in individuals with IHD. Low levels of PA independently contribute to increased death and adverse events in patients with IHD. Rates of PA in IHD patients continue to be unacceptably low in both hospital-based cardiac rehabilitation and home settings. Compounding this issue is often the symptom of hopelessness. The links among hopelessness, PA and mortality and morbidity for patients with IHD remain largely unknown, especially in rural and minority IHD patients. The purpose of this study is to delineate differences in hopelessness between urban and rural patients with IHD, as well as between racial minority, including Hispanic and Native American, and White patients with IHD. Potential mediation of urbanicity and race/ethnicity by social connectedness, a key variable in rural settings, will also be examined. A 6-month longitudinal study will be conducted at Sanford Heart Hospital and Avera Health in Sioux Falls, South Dakota. Hopelessness will be measured using the State-Trait Hopelessness Scale. The results of this study have potential to transform nursing practice by providing a better understanding of hopelessness in IHD patients and informing future exercise rehabilitation studies and interventions in rural and minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction or unstable angina or having undergone a percutaneous coronary intervention or coronary artery bypass surgery
* ≥ 18 years
* planned discharge home
* cognitive and physical ability to complete the study measures.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized individuals
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
State and Trait levels of Hopelessness | Six-month
  State-Trait Hopelessness Scale (values range from 1-4 on both subscales with larger values meaning more hopelessness)

SECONDARY OUTCOMES:
Participation (yes/no) and Levels (frequency; vigor) of Exercise | Six-month
  CREPT measurement tool for self-reported home and hospital exercise participation (yes/no) and levels (frequency/vigor) of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Tintle, Principal Investigator — Dordt University
Locations (2):
- United States (2):
  - Avera Health, Sioux Falls, South Dakota
  - Sanford Health, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bomgaars D, Jensen GA, White LL, Van De Griend KM, Visser AK, Goodyke MP, Luong A, Tintle NL, Dunn SL. Investigating Rurality as a Risk Factor for State and Trait Hopelessness in Hospitalized Patients With Ischemic Heart Disease. J Am Heart Assoc. 2021 Sep 7;10(17):e020768. doi: 10.1161/JAHA.121.020768. Epub 2021 Sep 1. PMID 34465185